IRB Approved: 16 Apr 2024 Version 1.0

# Evaluation of Wear Experience with PRECISION7® Contact lenses in habitual Acuvue® Oasys® lens wearers

**Protocol Number: 2024H0089** 

NCT Number: NCT06382064

Version 1.0

16 Apr 2024

Version 1.0

## Evaluation of Wear Experience with PRECISION7® Contact lenses in habitual Acuvue® Oasys® lens wearers

Jennifer Fogt, OD MS

The Ohio State University College of Optometry
Innovation in Vision and Eye care Research Group - iVERG
338 West 10<sup>th</sup> Ave
Columbus OH 43210
Phone: 614-292-0882

## **Purpose**

The purpose of this study is to explore the wear experience of current Acuvue Oasys lens wearers after they have been fit into PRECISION7® Contact Lenses.

## **Study Overview**

This open-label study is of current Acuvue® Oasys® wearers (2 – week replacement, reusable lenses) who are satisfied with their current lenses. Subjects will be refit into PRECISION7® contact lenses and will wear lenses for approximately 2 weeks. Subjects will return for vision and lens fit assessments and will complete surveys about their wear experience.

## **Background**

Soft daily wear contact lenses are used by an estimated 40.9 million adults in the United States.<sup>1</sup> Contact lenses which are worn for daily wear are considered minimal risk by the FDA, and risks to wearers are minimized by proper lens care and hygiene. The subjects in this study are current satisfied wearers of 2 week planned replacement lenses (Acuvue® Oasys®) and will be fit into PRECISION7® 1 week reusable contact lenses.

## **Key Endpoint:**

Subjective assessment of P7 experience with CLDEQ-8

## **Exploratory Endpoints:**

- Visual Analog Scale survey of lens wear symptoms (comfort, dryness, vision, satisfaction)
- Assessment via questionnaire about quality of life, preference, and lens modality experience

## **Study Time Points:**

Version 1.0

After responding to recruitment material, potential participants will respond to pre-screening questions to determine initial eligibility. Those eligible will be scheduled for a screening visit and will complete the informed consent process. Participants should report to the exam wearing existing current Acuvue® Oasys® lenses with a copy of their current prescription or packaging. Visual acuity and an evaluation of the subject's ocular health will occur to determine eligibility including positively responding to the question, "Are you satisfied with your current Acuvue Oasys contact lenses?" Acuvue Oasys lenses will be evaluated and optimized before dispensing a new pair of lenses for 2 weeks of wear (-3 days). Assessments of initial satisfaction, initial comfort, and initial vision will also be complete.

Visit 2: Acuvue Oasys contact lens follow up and Precision 1 fitting visit. Patients will be asked if they are still satisfied with their current Acuvue® Oasys® contact lenses in order to proceed and vision, lens fit and ocular health will be assessed. Subjects will then be fit with PRECISION7® Contact Lenses with assessments of initial satisfaction, initial comfort, and initial vision. Lenses will be dispensed and a contact lens follow-up visit will be scheduled for 2 weeks (-3 days)

**Visit 3: The contact lens follow up visit** will occur approximately 2 weeks (-3 days) following the initial fitting. Subjects will have visual acuity, an assessment of ocular health, and lens fit completed. Subjects will then complete surveys about their lens wear experience.

## All surveys will be completed in REDCap.<sup>2,3</sup>

## Surveys will include:

CLDEQ-8

Initial impression VAS surveys

Initial vision

Initial comfort

Initial satisfaction

VAS survey of comfort/dryness/vision

0-100 scale:

Overall Quality of vision

End of Day Quality of vision

Overall comfort

End of Day comfort

Overall dryness

End of Day dryness

Overall satisfaction

End of Study Wear Experience

Convenience of 1 week replacement lens, preference for 1 week replacement lens, ease of use

Would you purchase/switch to P7?

Satisfaction with P7

## Quality of Life

Quality of vision while watching television, using your smart phone, dining out, working out, reading a book/magazine/newspaper

Comfort while watching television, using your smart phone, dining out, working

Version 1.0

## out, reading a book/magazine/newspaper

#### Recruitment

Potential subjects may see posters placed on bulletin boards locally, at The Ohio State University, or local eye care offices, student dorms, emails to students, faculty and staff at OSU, online or paper ads, or signs on the OSU buses. Facebook advertising through the CCTS will occur. A search of the electronic medical records of The Ohio State College of Optometry may be done to identify possible subjects who then may be contacted by email or phone with information about the study. Word of mouth referrals by study team members to OSU employees and friends may occur. Emails to alumni of the OSU College of Optometry may be sent for local doctors to notify eligible potential subjects about the study.

## Inclusion criteria:

- Subjects must be current Acuvue® Oasys® spherical lens wearers.
- Subjects must have 20/25 or better distance visual acuity with current lenses in each eye.
- Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI)
- Ability to give informed consent
- Willing to spend time for the study. Subjects will be required to attend three study visits and wear contact lenses on days between study visits.
- Either gender
- Any racial or ethnic origin

#### **Exclusion criteria:**

- Current ocular inflammation or infection as assessed by the study investigator
- Currently pregnant or lactating.
- Systemic inflammatory disease (i.e. Diabetes, etc.) that could confound study results in the opinion of the investigator

## **Consent and Confidentiality**

A team member trained in the consent process will provide the consent document for the potential subject to read and will review the procedures with reference to the consent form. The individual is then provided with time to read the consent form and offered the opportunity to ask questions. The participant is explicitly told that they may stop participation at any time. All subjects will have the capacity to give informed consent. If there is any doubt as to the subject's ability to consent to the study, the subject will be excluded from the study. If the subject agrees to take part in the screening or measurement, he or she will sign and date the most recent IRB-stamped consent as will the team member. The subject will be provided with a copy of the consent form.

Version 1.0

The investigator team is trained in privacy issues and will be reminded of the importance of patient privacy prior to study initiation. Potential study participants will contact us after seeing advertisements, emails or hearing about the study by word of mouth, giving them the choice of whether or not they wish to participate in a study for people with dry eyes. Privacy is protected by limiting information related to study recruitment only, and no other personal or medical information that should be private to the patients. The PHI needed is only for the purposes of this study. It is highly unlikely, indeed extremely remote that the dry eye symptoms or signs are related to private or personal information that should or would be preferred to be kept confidential to the patients. Risk factors for dry eye rarely relate to matters or conditions that would be personal to the patient such as personal relationships, behaviors or diseases that one prefers to keep private and confidential.

## **Statistical Analysis**

This pilot study was not intended (powered) to prove superiority, but to study the acceptability of the study lens in previous successful Acuvue® Oasys® wearers. The study reported outcomes using descriptive statistics, and as such, no power calculation was necessary. Several contact lens studies have been conducted at this site which successfully recruited 50 participants. Eighty potential participants will be screened in order to complete 60 participants.

## **Data Management and Security**

During the active stages of the study (recruitment to last measurement visit), all paperwork (consents, questionnaires and data forms) for each subject will reside in a subject folder for easy access throughout the study. The folders will reside in the limited-access research area, in a locked file drawer or cupboard. At the completion of the study or disenrollment of a subject the paperwork in the subject's folders will be reorganized into a regulatory binder (consents, W-9s) and a data binder (questionnaire and data forms) and will reside in an office in the limited-access research area. When the data analysis is completed and the study is considered complete, the binders will be stored in the secure Department or Office Clinical Research Area. Paperwork (questionnaire and data forms) for individuals who participate in the baseline visit but are not eligible to continue the study will be stored in the study regulatory binder in an office in the limited-access research area. An electronic file of potential subjects and a file of enrolled subjects with their contact information, as well as electronic files of collected data with the subject number, will reside on a limited-access shared drive with firewall and password protection and is restricted to individuals in the research team. Any electronic data files that contain PHI will be destroyed at the conclusion of the study.

## **Risks to Subjects and Mitigation**

Although rare, a subject could experience eye pain, changes in vision, continued redness or irritation of the eye when inserting or learning to insert a contact lens. More likely transient blurring of vision (less than one minute) or mild, transient (less than a minute) stinging may occur.

Version 1.0

#### **Adverse Events**

All adverse events will be documented and reported under the guidelines of The Ohio State University Event Reporting guidelines, with any serious, unanticipated and related events being reported to the IRB, by the PI, within 10 days. Adverse Events information will be summarized in the annual report to the IRB at the end of the study. Adverse events will be assessed and determined by Dr. Jennifer Fogt.

## **Subject Dismissal**

Subjects who, after study team member coaching, are not able to provide analyzable data may be dismissed from the study. Analyzable data is, for example, that which is obtained for the entire measurement interval and provides a readable eye image. Data may not be analyzable if patient isn't able to stand or move freely to utilize the equipment, to name just two causes issues. These issues are usually revealed at the screening assessment visit. Subjects who cannot provide analyzable data will be dismissed for the study. Subjects who do not keep scheduled visits within the required time frame will be dismissed from the study. Study team members will make reasonable efforts to accommodate subjects' schedules.

#### **Protocol Violations, Discontinuation**

In the event that a member of the study team or a representative of sponsor becomes aware of a major protocol violation, the IRB shall be notified within 10 working days.

## References

- 1. Cope JR, Collier SA, Rao MM, et al. Contact Lens Wearer Demographics and Risk Behaviors for Contact Lens-Related Eye Infections--United States, 2014. *MMWR Morb Mortal Wkly Rep.* 2015;64(32):865-870.
- 2. Harris PA, Taylor R, Minor BL, et al. The REDCap consortium: Building an international community of software platform partners. *J Biomed Inform.* 2019;95:103208.
- 3. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)-A metadata-driven methodology and workflow process for providing translational research informatics support. *J Biomed Inform.* 2009;42(2):377-381.